CLINICAL TRIAL: NCT06592469
Title: The Outcome of Ureteroscopy in Fresh Versus Recurrent Cases of Stone Ureter (Post-ESWL, Endoscopy, or Open Surgery)
Brief Title: Outcome of URS in Fresh Versus Recurrent Cases of Stone Ureter
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Moustafa Hussein Soliman, Resident doctor, Assiut University
Other Study IDs: Outcome of Ureteroscopy
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stone Ureter
Keywords: URS
MeSH Terms: conditions — Ureterolithiasis | interventions — Ureteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fresh cases: Outcome of URS in fresh stone ureter
  Interventions: Procedure: Ureteroscopy
- Recurrent cases: Outcome of URS in recurrent cases of stone ureter post ESWL ,URS , open surgery
  Interventions: Procedure: Ureteroscopy

INTERVENTIONS:
Procedure: Ureteroscopy — URS is done to each group to reveal outcome of stone free rate in fresh versus recurrent cases of stone ureter
  Other Names: URS

SUMMARY:
Comparison of Ureteroscopy in fresh versus recurrent cases of stone ureter

DETAILED DESCRIPTION:
Urolithiasis is a common cause of both urology outpatient clinic and emergency room encounters. Approximately 75-90% of ureteral stones pass spontaneously. from this point of view other managements of ureteric stones either ESWL, ureteroscopy or open surgery according to location, site, size, and density. Ureteroscopy is commonly used to diagnose and treat kidney and ureteral stones, ureteral strictures, and urothelial cancers. Semirigid URS is the gold standard of treatment for ureteral stones. High success rates and low morbidity have been reported in semirigid URS. but complications still occur in some cases. The possibility to predict their occurrence should influence patient advisement and better case selection. there are many predictors of successful URS as age, gender, previous ESWL, and stone character. In addition, the impacted stone is a risk factor, and it is described in the literature as ureteral wall thickness, higher grades of hydronephrosis, ureteral stricture, polyp, inflammatory reaction, and difficulty to introduce the guide wire. the literature is very poor in illustrating the previous procedures as a predictor of successful URS only seen in very few original articles as second-time URS after any procedure decreases the rate of success, so it is a point of research that Amr Moustafa aims to clarify. Amr Moustafa will conduct a prospective study to evaluate the outcomes of URS for stones in the fresh and recurrent cases.

ELIGIBILITY:
Inclusion Criteria:

* • all cases with middle and lower ureteric stone candidate for endoscopy.

  * Stone 15mm or less.

Exclusion Criteria:

* • Patients with a ureteral stent.

  * Patient refusing participation.
  * Pregnant woman.
  * Active urinary tract infection.
  * Comorbidities prevent intervention including bleeding tendency or uncorrectable coagulation profile.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: .4. 2- Study subjects:
  1. Inclusion criteria:
     * all cases with middle and lower ureteric stone candidate for endoscopy.
     * Stone 15mm or less.
  2. Exclusion criteria:
     * Patients with a ureteral stent.
     * Patient refusing participation.
     * Pregnant woman.
     * Active urinary tract infection.
     * Comorbidities prevent intervention including bleeding tendency or uncorrectable coagulation profile.
  3. Sample Size Calculation:
  Based on previously reported frequency of primary failure of ureteocopy in case of recurrent stone that ranged between 1-37% (*reference)* a total sample size of 62 patients will be required ( 31 patients in each arm) with the following assumption; alpha error 5%, 80% power with 95% confidence interval
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Stone free rate of Urereroscopy in fresh versus recurrent cases of stone ureter | 1 day post operative by MSCTKUB or Plain KUB to determine residual stones post operative
  • Stone free rate with a mean operative time of 1 hr by MSCTKUB or Plain KUB to determine residual stones post operative

SECONDARY OUTCOMES:
• Rate of intraoperative findings in each group. | Intraoperative
  • Rate intraoperative findings in each group by ureteroscope
• The rate of complication in each group | Intraoperative by ureteroscope and one day post operative by MSCT
  To determine rate of intraoperative complications as bleeding , ureteric perforation , residual stones
• The rate of stone impaction in each group | Intraoperative by ureteroscope
  Rate of stone impaction in each group fresh and recurrent cases

CONTACTS AND LOCATIONS:
Overall Officials: Fathy Gaber Mahmoud Alanany, Prof of URO, Study Director — Assiut University; Mahmoud M. Shalaby, Prof of URO, Study Director — Assiut University; Nasreldin Abdeal Mohammed, Ass Prof, Study Director — Assiut University
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Egypt

REFERENCES:
- See also: Factors predicting duration and success of semirigid ureteroscopy for ureteral stones in different localizations — https://pubmed.ncbi.nlm.nih.gov/33818430/
- See also: Assessment of factors affecting the spontaneous passage of lower ureteric calculus on the basis of lower ureteric calculus diameter, density, and plasma C-reactive protein level. Urology Annal — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6060607/
- See also: Stone composition independently predicts stone size in 18,029 spontaneously passed stones — https://pubmed.ncbi.nlm.nih.gov/30719571/
- See also: Outcomes of Shock Wave Lithotripsy and Ureteroscopy for Treatment of Pediatric Urolithiasis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6103480/
- See also: Pushing the boundaries of ureteroscopy: current status and future perspectives — https://pubmed.ncbi.nlm.nih.gov/24890883/
- See also: Semirigid Ureteroscopy: Step by Step — https://pubmed.ncbi.nlm.nih.gov/32459149/
- See also: Complications of pneumatic ureterolithotripsy in the early postoperative period — https://pubmed.ncbi.nlm.nih.gov/15735383/
- See also: Complications of 2735 retrograde semirigid ureteroscopy procedures: a single-center experience — https://pubmed.ncbi.nlm.nih.gov/16548724/
- See also: Endoscopic features of impacted ureteral stones — https://pubmed.ncbi.nlm.nih.gov/14665851/
- See also: Predictive factors for intraoperative complications in semirigid ureteroscopy: analysis of 1235 ballistic ureterolithotripsies — https://pubmed.ncbi.nlm.nih.gov/18632141/
- See also: Revisiting the predictive factors for intra-operative complications of rigid ureteroscopy: a 15-year experience — https://pubmed.ncbi.nlm.nih.gov/22641488/